CLINICAL TRIAL: NCT06049368
Title: 68Ga-P16-093 PET/CT Imaging in the Salivary Gland
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-PSS093
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Primary Sjögren Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-P16-093 (Experimental): Within 1 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-P16-093.
  Interventions: Drug: 68Ga-P16-093

INTERVENTIONS:
Drug: 68Ga-P16-093 — Intravenous injection of 68Ga-P16-093 with the dosage of 1.5-1.8 MBq (0.04-0.05 mCi)/kg. Tracer doses of 68Ga-P16-093 will be used to image lesions of glioma by PET/CT.

SUMMARY:
Prostate specific membrane antigen (PSMA) is a type II transmembrane protein and acts as a glutamate carboxypeptidase enzyme. It is first described in prostate cancer cell lines and later identified in various tissues, include salivary gland. This pilot study was designed to evaluate the diagnostic performance of 68Ga-P16-093 in primary sjogren's syndrome patients.

DETAILED DESCRIPTION:
Primary sjogren's syndrome (pSS) is a systemic autoimmune disease mainly presented hyperglobulinemia and exocrine gland involvement,and lack of diagnostic gold standard.Prostate-specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. However, PSMA is also expressed by various solid organs , such as salivary gland,which is often observed damage in primary Sjogren's syndrome patients.Therefore, PSMA may be an ideal target for evaluating salivary gland injury.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis confirmed by operation or biopsy.
* Obtain written informed consent and accepted follow-up.

Exclusion Criteria:

* Pregnant, lactating women or having parenting plans during the study
* Head and neck radiotherapy history ;
* Active hepatitis C infection (PCR positive), include immunodeficiency syndrome, sarcoidosis, amyloidosis, graft versus host disease, IgG4 related diseases.
* Other situaition researchers considered it was not appropriate to participate in trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | through study completion, an average of 1 year
  evaluating the number of regions in damaged salivary glands detected by 68Ga-P16-093

SECONDARY OUTCOMES:
standardized uptake value (SUV) of lesion | through study completion, an average of 1 year]
  comparing the SUVmax of different grades in salivary gland lesion, derived from 68Ga-P16-093

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital